CLINICAL TRIAL: NCT02399579
Title: Evaluation of a New Self-Assessed, Home-Based Symptom Score Test in Cat Allergic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: ZU-HypoScore-001
Record Dates: First submitted 2015-03-17; First posted 2015-03-26 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-07

CONDITIONS: Cat Allergy
Keywords: cat allergy; symptom score

ARMS (1):
- HypoScore (Experimental): Provocation test. Recording symptoms of cat allergic participants with the cat owner's cat: Before and after petting the cat.
  Interventions: Other: Provocation test

INTERVENTIONS:
Other: Provocation test — The participants will perform 8 provocation tests. Every provocation test consists of petting the cat until the participants become symptomatic. The symptoms of cat allergic participants with the cat owner's cat will be recorded before and after petting the cat.

SUMMARY:
The purpose of this study is to better standardize the symptom recording of cat allergic persons under real-life conditions. A new self-assessed, home-based symptom score will be tested.

DETAILED DESCRIPTION:
In order to bring research on cat dander allergy a step further we aim to investigate cat dander allergy symptoms and record them in a natural environment, respectively, i.e. at the participant's home. For this purpose we aim to test a new self-assessed, homebased symptom score (called HypoScore). The participants will perform 8 provocation tests. Every provocation test consists of petting the cat until the participants become symptomatic. The participants have to pet the cat everytime in the same manner. Directly before and after the provocation test the symptoms will be recorded in the eCRF by using an iPad mini.

ELIGIBILITY:
Inclusion Criteria:

* Participant understands the nature, meaning and scope of the study.
* Signed Informed Consent after being informed.
* Male and Female patients 18 years to 65 years of age.
* Positive screening prick test (mean wheal diameter ≥ 3 mm) when tested with already standardized cat allergen extract.
* Positive screening prick test (wheal diameter ≥ 3mm) to Histamine dihydrochloride 10mg/ml.
* Positive Scratch Test when tested with cat dander sample of participant's cat.
* Baseline symptoms with a severity of at least "1" in minimal 2 various symptoms.
* Owner of a cat that lives in the same household.

Exclusion Criteria:

* Impaired in understanding the nature, meaning and scope of the study or incapable of giving written informed consent
* Participation in another study with investigational drug within the 30 days preceding and during the present study
* Women who are pregnant or breast feeding
* Intention to become pregnant during the course of the study
* Positive skin reaction in the prick test to negative control
* History of anaphylactic reaction to pet allergens
* Severe diseases influencing the results of the present study by discretion of the investigator
* Immunotherapy with fel d 1 / cat allergen preparation during the past two years
* Skin lesions and excessive hair-growth in the skin test areas
* Treatment with prohibited concomitant medications with the exception of medications with local effects which will not influence the results of the skin tests and the results of the other tests (testing period).
* The patient should not suffer from other respiratory allergies during this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Time until the participant becomes symptomatic | approx. 15 minutes (during Provocation Test)
  How long can the owner pet his/her cat until he becomes symptomatic?

SECONDARY OUTCOMES:
Number of score points resulting from symptom score recording before and after the provocation test. | approx. 15 minutes (before and after provocation)
Visual Analogue Scale Values | approx. 5 minutes (before provocation)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M. Kündig, PD Dr. med., Principal Investigator — University of Zurich
Locations (1):
- Clinical Trial Center of the University Hospital Zurich, Zurich, Canton of Zurich, Switzerland